CLINICAL TRIAL: NCT02445976
Title: A Phase 2 Open-label Study to Evaluate the Efficacy and Safety of Seviteronel in Subjects With Castration-Resistant Prostate Cancer Progressing on Enzalutamide or Abiraterone
Brief Title: Once-daily Oral Seviteronel in Patients With Castration-Resistant Prostate Cancer Progressing on Enzalutamide or Abiraterone.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innocrin Pharmaceutical (Industry)
Collaborators: Prostate Cancer Foundation (Other); Prostate Cancer Clinical Trials Consortium (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INO-VT-464-CL-003; VMT-VT-464-CL-003 (Other: Innocrin)
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Prostate Cancer
Keywords: mCRPC; metastatic; castration-resistant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — seviteronel

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prior Abiraterone or Enzalutamide (Experimental): Seviteronel: given orally once daily in 28-day cycles
  Interventions: Drug: Seviteronel: given orally once daily in 28-day cycles
- Prior Abiraterone and Enzalutamide (Experimental): Seviteronel: given orally once daily in 28-day cycles
  Interventions: Drug: Seviteronel: given orally once daily in 28-day cycles

INTERVENTIONS:
Drug: Seviteronel: given orally once daily in 28-day cycles — Oral Seviteronel given once daily, in continuous 28-day cycles at the recommended Phase 2 dose
  Other Names: Seviteronel

SUMMARY:
The goal of this clinical study is to determine the efficacy and safety of Seviteronel, a lyase-selective inhibitor of CYP17 and an androgen receptor antagonist, in patients with castration-resistant prostate cancer (CRPC) who have been previously treated with enzalutamide and/or abiraterone.

DETAILED DESCRIPTION:
This is a phase 2 clinical trial of Seviteronel (an oral, potent and lyase-selective CYP17 inhibitor) in men with castration-resistant prostate cancer (CRPC) progressing on enzalutamide or abiraterone. Approximately 197 subjects will be used to assess treatment efficacy. The study will be conducted in two different clinical cohorts separated by prior exposure to enzalutamide or abiraterone, or prior exposure to enzalutamide and abiraterone.

ELIGIBILITY:
Inclusion Criteria

1. Subjects must be ≥18 years of age.
2. Subjects or their legal representatives must be able to provide written informed consent.
3. Subjects must have documented histological or cytological evidence of adenocarcinoma of the prostate.
4. Subjects must have an ECOG Performance Score of 0-1.
5. Subjects must have undergone orchiectomy, or have ongoing LHRH analogue therapy prior to drug initiation. Subjects on LHRH analogues must remain on these agents for the duration of the study.
6. Subjects must have castrate levels of testosterone (≤50 ng/dl [1.7 nmol/L]) and have progressive disease at Screening defined as PSA rise determined by a minimum of 2 rising PSA values ≥1 week between each assessment. The PSA value at the Screening visit must be ≥2ng/mL with or without:

   * Soft tissue disease progression defined by RECIST 1.1 at Screening or ≤ 28 days of C1D1. Measurable disease is not required for entry. Lymph nodes ≥ 1.5cm (short axis) are considered measurable disease (PCWG3)
   * Bone disease progression defined by ≥2 new lesions on bone scan at Screening, or ≤28 days of C1D1
7. Subjects must have received abiraterone and/or enzalutamide. Subject must have received either abiraterone or enzalutamide for ≥12 weeks. Other second generation CYP17 inhibitors/androgen receptor antagonists including but not limited to TAK-700 (orteronel), TOK-001 (galeterone) may have been taken in place of abiraterone and ARN-509 (apalutamide) may have been taken in place of enzalutamide.
8. Subjects must have adequate hematopoietic function as evidenced by:

   * WBC ≥3,000/µl
   * ANC ≥1,500/µl
   * Platelet count ≥100,000/µl
   * HGB ≥10 g/dl and not transfusion dependent
9. Subjects must have adequate liver function, including all of the following:

   * Total serum bilirubin ≤2.0 x ULN unless the subject has documented Gilbert syndrome;
   * Aspartate and alanine aminotransferase (AST & ALT) ≤3.0 x ULN or ≤5.0 x ULN if subject has liver metastasis;
   * Alkaline phosphatase ≤2.0 x ULN or ≤5 x ULN in case of bone metastasis and/or hepatic metastasis
10. Subjects must have adequate renal function as evidenced by a serum creatinine of <2.0 mg/dl.
11. Subjects must have potassium (K+) >3.5 mEq/l.
12. Subject and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (one of which must include a condom as a barrier method of contraception) starting a Screening and continuing throughout the study period and for 3 months after final study drug administration • Two acceptable forms of birth control include:

1. Condom (barrier method of contraception), and 2. One of the following:

1. Oral, injected or implanted hormonal contraception
2. Placement of an intrauterine device (IUD) or intrauterine system (ISU)
3. Additional barrier methods of contraception: Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
4. Vasectomy or surgical castration ≥ 6 months prior to Screening. 13. Subjects able to swallow study medication 14. Subjects able to comply with study requirements

Exclusion Criteria

1. Subjects who have completed sipuleucel-T (Provenge ®) treatment within 28 days of study drug initiation.
2. Subjects on 5-alpha reductase inhibitors such as finasteride (PROSCAR®, PROPECIA®), or dutasteride (AVODART®) within 28 days of study drug initiation.
3. Subjects who received any investigational agent ≤28 days of study drug initiation.
4. Subjects who received palliative radiotherapy ≤2 weeks of study drug initiation.
5. Subjects with symptomatic CNS metastases.
6. Subjects with a history of another invasive malignancy ≤3 years of study drug initiation.
7. Subjects with a QTcF interval of >470 msec; if the Screening ECG QTcF interval is >470 msec, it may be repeated, and if repeat <470 msec, the subject may be enrolled.
8. Subject with clinically significant cardiac arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes, second degree or third degree atrioventricular heart block without a permanent pacemaker in place)
9. Subject that started a bone modifying agent (e.g. bisphosphonates, denosumab) ≤ 28 days of study drug initiation (note: ongoing bone modifying agents administered > 28 days are allowed).
10. Subject with any medical condition that could preclude subject participation in the study, pose an undue medical hazard, or which could interfere with study results.
11. Subject with Class III or IV Congestive Heart Failure as defined by the New York Heart Association (NYHA) functional classification system within the previous 6 months.
12. Subject with a history of loss of consciousness or transient ischemic attack ≤ 12 months of study drug initiation.
13. Subject with known active HIV, Hepatitis B, or Hepatitis C infections.
14. Subject with known or suspected hypersensitivity to seviteronel, or any components of the formulation
15. Subject with any other condition which in the opinion of the investigator would preclude participation in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-12 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who have a PSA response by while on study from starting treatment with seviteronel | 6 months
  PSA response at any time whilst on study from the start of treatment within seviteronel defined by a ≥ 50% decrease in serum PSA.
The time to radiographic disease progression by RECIST 1.1 or PCWG3 | 10 months
  Median time to radiographic disease progression evaluated by computerized tomography (CT scan) or magnetic resonance imaging (MRI) and radionuclide bone scans by RECIST 1.1 or Prostate Cancer Clinical Trials Working Group 3 (PCWG3)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - University of Alabama, Birmingham, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - University of California at Los Angeles, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Tulane University, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - GU Research Network, Omaha, Nebraska
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - University of Virginia, Charlottesville, Virginia
  - Virginia Oncology Associates, Hampton, Virginia
  - University of Washington, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin